CLINICAL TRIAL: NCT03455608
Title: PRO-ACTIVE: Comparing The Effectiveness of Prophylactic Swallow Intervention for Patients Receiving Radiotherapy for Head and Neck Cancer
Brief Title: PRO-ACTIVE: Prophylactic Swallow Intervention for Patients Receiving Radiotherapy for Head and Neck Cancer
Acronym: PRO-ACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Applied Health Research Centre (Other); Qualitative Health Research Consultants, LLC (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO1363
Record Dates: First submitted 2018-02-11; First posted 2018-03-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Dysphagia
Keywords: dysphagia; swallowing disorder; speech pathology; swallowing therapy; head and neck cancer; radiotherapy; toxicity; supportive care
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RE-ACTIVE (Active Comparator): Reactive intervention started promptly if/when dysphagia is identified (RE-ACTIVE)
  Interventions: Behavioral: RE-ACTIVE
- PRO-ACTIVE EAT (Active Comparator): Early low intensity proactive intervention started before RT commences
  Interventions: Behavioral: PRO-ACTIVE EAT
- PRO-ACTIVE EAT + EXERCISE (Active Comparator): Early high intensity proactive intervention started before RT commences
  Interventions: Behavioral: PRO-ACTIVE EAT + EXERCISE

INTERVENTIONS:
Behavioral: RE-ACTIVE — Reactive intervention started promptly if/when dysphagia is identified
  Arms: RE-ACTIVE
Behavioral: PRO-ACTIVE EAT — Early low intensity proactive intervention started before RT commences
  Arms: PRO-ACTIVE EAT
Behavioral: PRO-ACTIVE EAT + EXERCISE — Early high intensity proactive intervention started before RT commences
  Arms: PRO-ACTIVE EAT + EXERCISE

SUMMARY:
Dysphagia (difficulty swallowing) is a common and potentially life-threatening toxicity of radiotherapy (RT) for patients with head and neck cancer (HNC). HNC survivors have a 20-24 percent lifetime risk of pneumonia after RT, which is associated with a 42 percent excess risk of death in survivorship. Moreover, dysphagia predisposes individuals to malnutrition, and at least half of HNC patients require feeding tubes during RT.

Patients are commonly referred for swallowing therapy with a speech pathologist. Some patients receive early intervention, before a swallowing problem begins-PRO-ACTIVE therapy. Other patients are monitored and prescribed dysphagia interventions only if and when a swallowing problem occurs-RE-ACTIVE therapy. Thus, REACTIVE therapy aims to reverse an already impaired swallowing ability, whereas PRO-ACTIVE therapy aims to prevent or reduce severity of dysphagia. These two broad categories of therapy represent the most common types of intervention offered to HNC patients across North America. Although there is single-institution evidence to support each practice, it is yet unknown which is most effective.

To address this gap, the primary aim of this international, multi-site 3-arm pragmatic randomized clinical trial is to compare the effectiveness of PRO-ACTIVE (high and low intensity) versus RE-ACTIVE swallowing therapy among 952 patients with HNC planning to undergo RT, using duration of feeding tube dependence after RT as the primary outcome. Our secondary aim proposes to compare the relative benefit or harm of these swallowing interventions on secondary outcomes considered relevant to our stakeholder partners.

DETAILED DESCRIPTION:
Swallowing therapy is commonly provided as a behavioral treatment to lessen the risk or severity of dysphagia in head and neck cancer (HNC) patients; however, best practice is not established. This multi-site, international randomized clinical trial (RCT) will compare the effectiveness of PRO-ACTIVE (high and low intensity) versus RE-ACTIVE swallowing interventions in 952 HNC patients undergoing radiotherapy (RT). The 3 study arms represent alternate timing and intensity of swallowing therapy delivered by a speech language pathologist: 1) RE-ACTIVE, 2) PRO-ACTIVE EAT, and 3) PRO-ACTIVE EAT + EXERCISE.

The primary aim of the PRO-ACTIVE trial is to compare the effectiveness of PRO-ACTIVE versus RE-ACTIVE swallowing interventions among patients with HNC planned to undergo RT. We hypothesize that the combined PRO-ACTIVE therapies are more effective than RE-ACTIVE therapy; and, if so, that more intensive PRO-ACTIVE (EAT + EXERCISE) is superior to less intensive PRO-ACTIVE (EAT). Effectiveness will be measured based on reduced duration of feeding tube dependency as the primary endpoint, an outcome valued equally by patients, caregivers and clinicians.

The secondary aim of the PRO-ACTIVE trial is to compare the relative benefit or harm of swallowing therapy arms on secondary outcomes including videofluoroscopic swallowing evaluations, functional status measures, health status measures, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age diagnosed with head and neck malignancy;
* RT treatment planned for curative intent;
* Dispositioned to receive external beam radiotherapy dose ≥60 gray to bilateral fields at participating institution;
* Sufficient fluency in written English, French, Spanish or Simplified Chinese to be able to complete the study patient reported outcome questionnaires

Exclusion Criteria:

* Distant metastasis at enrollment; or
* Prior or planned total laryngectomy; or
* Moderate/severe dysphagia at enrollment per baseline videofluoroscopy DIGEST grade ≥2 (as graded per central laboratory review)
* Previously seen by speech language pathologist for swallowing therapy for the current head and neck cancer
* Diagnosis of second primary non-head and neck cancers in the thorax or the central nervous system at enrollment
* Head and neck radiotherapy for thyroid or cutaneous/skin primary tumors, regardless of neck fields

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Duration of feeding tube dependence | Baseline - 12 months
  Effectiveness will be measured based on duration of feeding tube dependency (count of days from end of radiotherapy to last feeding tube use within the 12-month study period)

SECONDARY OUTCOMES:
The MD Anderson Dysphagia Inventory (MDADI) | Baseline, Week 6/7, 3 months, 12 months
  Measurement of swallowing-related Quality of Life
The MD Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) | Baseline, Week 2, Week 4, Week 6/7, 3 months, 12 months
  Measurement of severity or burden of cancer-related symptoms and interference with daily functioning.
Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) | Baseline, 3 months, 12 months
  Videofluoroscopy study score ranging from 0 to 5, where 4 is worst.
Pharyngeal Constriction Ratio (PCR) | Baseline, 3 months, 12 months
  Videofluoroscopy study score ranging from 0 to 1, where 1 is worst.
Penetration-Aspiration Scale (PAS) | Baseline, 3 months, 12 months
  Videofluoroscopy study score ranging from 1 to 8, where 8 is worst.
Peak esophageal opening | Baseline, 3 months, 12 months
  Videofluoroscopy study score ranging from 0 to infinity, where lower value is worse.
Performance Status Scale Head and Neck (PSS-HN) | Baseline, Week 2, Week 4, Week 6/7, 3 months, 12 months
  Measurement of swallowing and speech performance
Medical Outcome of Dysphagia (MOD) | Baseline, 3 months, 12 months
  Patient reported symptoms related to health consequences secondary to dysphagia, namely: malnutrition, aspiration pneumonia and mood changes such as depression and anxiety
Cancer Behavior Inventory (CBI-V3) | Baseline, 3 months, 12 months
  Measurement of self-efficacy strategies for coping with cancer
EQ-5D-5L | Baseline, 3 months, 12 months
  Measurement of generic quality of life
Medical History | Baseline, Week 6/7, 3 months, 12 months
  Intake details, radiation therapy details, chemotherapy details, tumour status, surgery history, tracheotomy, feeding tube status, feeding tube dependence, concomitant therapies, and complication details.
Pain Medications | Baseline; Week 6/7, 3 Month, and 12 Months
  All pain medications (including over-the-counter) taken in the past 48 hours
Mouth Opening/Trismus | Baseline; 3 Month and 12 Months
  Measurement of interincisal opening
Hospitalization/Emergency Department (ED) Presentation | Baseline, Week 6/7, 3 months, 12 months
  Hospitalization/ED presentation at cancer hospital or any external institutions

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Martino, PhD, Principal Investigator — University Health Network, Toronto; Kate Hutcheson, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (13):
- United States (10):
  - University of Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krisciunas GP, Sokoloff W, Stepas K, Langmore SE. Survey of usual practice: dysphagia therapy in head and neck cancer patients. Dysphagia. 2012 Dec;27(4):538-49. doi: 10.1007/s00455-012-9404-2. Epub 2012 Mar 29. PMID 22456699
- [Background] Xu B, Boero IJ, Hwang L, Le QT, Moiseenko V, Sanghvi PR, Cohen EE, Mell LK, Murphy JD. Aspiration pneumonia after concurrent chemoradiotherapy for head and neck cancer. Cancer. 2015 Apr 15;121(8):1303-11. doi: 10.1002/cncr.29207. Epub 2014 Dec 23. PMID 25537836
- [Background] Hunter KU, Lee OE, Lyden TH, Haxer MJ, Feng FY, Schipper M, Worden F, Prince ME, McLean SA, Wolf GT, Bradford CR, Chepeha DB, Eisbruch A. Aspiration pneumonia after chemo-intensity-modulated radiation therapy of oropharyngeal carcinoma and its clinical and dysphagia-related predictors. Head Neck. 2014 Jan;36(1):120-5. doi: 10.1002/hed.23275. Epub 2013 Jun 1. PMID 23729173
- [Background] Hutcheson KA, Bhayani MK, Beadle BM, Gold KA, Shinn EH, Lai SY, Lewin J. Eat and exercise during radiotherapy or chemoradiotherapy for pharyngeal cancers: use it or lose it. JAMA Otolaryngol Head Neck Surg. 2013 Nov;139(11):1127-34. doi: 10.1001/jamaoto.2013.4715. PMID 24051544
- [Background] Setton J, Lee NY, Riaz N, Huang SH, Waldron J, O'Sullivan B, Zhang Z, Shi W, Rosenthal DI, Hutcheson KA, Garden AS. A multi-institution pooled analysis of gastrostomy tube dependence in patients with oropharyngeal cancer treated with definitive intensity-modulated radiotherapy. Cancer. 2015 Jan 15;121(2):294-301. doi: 10.1002/cncr.29022. Epub 2014 Oct 6. PMID 25286832
- [Background] Mortensen HR, Jensen K, Aksglaede K, Lambertsen K, Eriksen E, Grau C. Prophylactic Swallowing Exercises in Head and Neck Cancer Radiotherapy. Dysphagia. 2015 Jun;30(3):304-14. doi: 10.1007/s00455-015-9600-y. Epub 2015 Feb 19. PMID 25690840
- [Background] Ohba S, Yokoyama J, Kojima M, Fujimaki M, Anzai T, Komatsu H, Ikeda K. Significant preservation of swallowing function in chemoradiotherapy for advanced head and neck cancer by prophylactic swallowing exercise. Head Neck. 2016 Apr;38(4):517-21. doi: 10.1002/hed.23913. Epub 2015 Jun 16. PMID 25351675
- [Background] van der Molen L, van Rossum MA, Rasch CR, Smeele LE, Hilgers FJ. Two-year results of a prospective preventive swallowing rehabilitation trial in patients treated with chemoradiation for advanced head and neck cancer. Eur Arch Otorhinolaryngol. 2014 May;271(5):1257-70. doi: 10.1007/s00405-013-2640-8. Epub 2013 Jul 28. PMID 23892729
- [Background] Carroll WR, Locher JL, Canon CL, Bohannon IA, McColloch NL, Magnuson JS. Pretreatment swallowing exercises improve swallow function after chemoradiation. Laryngoscope. 2008 Jan;118(1):39-43. doi: 10.1097/MLG.0b013e31815659b0. PMID 17989581
- [Background] Shaw SM, Flowers H, O'Sullivan B, Hope A, Liu LW, Martino R. The effect of prophylactic percutaneous endoscopic gastrostomy (PEG) tube placement on swallowing and swallow-related outcomes in patients undergoing radiotherapy for head and neck cancer: a systematic review. Dysphagia. 2015 Apr;30(2):152-75. doi: 10.1007/s00455-014-9592-z. Epub 2015 Mar 4. PMID 25737196
- [Background] MD Anderson Head and Neck Cancer Symptom Working Group. Beyond mean pharyngeal constrictor dose for beam path toxicity in non-target swallowing muscles: Dose-volume correlates of chronic radiation-associated dysphagia (RAD) after oropharyngeal intensity modulated radiotherapy. Radiother Oncol. 2016 Feb;118(2):304-14. doi: 10.1016/j.radonc.2016.01.019. Epub 2016 Feb 17. PMID 26897515
- [Background] Eisbruch A, Kim HM, Feng FY, Lyden TH, Haxer MJ, Feng M, Worden FP, Bradford CR, Prince ME, Moyer JS, Wolf GT, Chepeha DB, Ten Haken RK. Chemo-IMRT of oropharyngeal cancer aiming to reduce dysphagia: swallowing organs late complication probabilities and dosimetric correlates. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):e93-9. doi: 10.1016/j.ijrobp.2010.12.067. Epub 2011 May 17. PMID 21592678
- [Background] Hutcheson KA, Lewin JS, Barringer DA, Lisec A, Gunn GB, Moore MW, Holsinger FC. Late dysphagia after radiotherapy-based treatment of head and neck cancer. Cancer. 2012 Dec 1;118(23):5793-9. doi: 10.1002/cncr.27631. Epub 2012 May 17. PMID 23640737
- [Background] Rubin EB, Buehler AE, Halpern SD. States Worse Than Death Among Hospitalized Patients With Serious Illnesses. JAMA Intern Med. 2016 Oct 1;176(10):1557-1559. doi: 10.1001/jamainternmed.2016.4362. No abstract available. PMID 27479808
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] National Cancer Institute. SEER cancer statistics factsheets: Larynx cancer. http://seer.cancer.gov/statfacts/html/laryn.html. Accessed December 12, 2016.
- [Background] Canadian Cancer Society's Advisory Committee on Cancer Statistics. Canadian cancer statistics 2016. 2016; http://www.cancer.ca/en/cancer-information/cancer-101/canadian-cancer-statistics-publication/?region=on. Accessed December 12, 2016.
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Weinberger PM, Yu Z, Haffty BG, Kowalski D, Harigopal M, Brandsma J, Sasaki C, Joe J, Camp RL, Rimm DL, Psyrri A. Molecular classification identifies a subset of human papillomavirus--associated oropharyngeal cancers with favorable prognosis. J Clin Oncol. 2006 Feb 10;24(5):736-47. doi: 10.1200/JCO.2004.00.3335. Epub 2006 Jan 9. PMID 16401683
- [Background] Roe JW, Carding PN, Rhys-Evans PH, Newbold KL, Harrington KJ, Nutting CM. Assessment and management of dysphagia in patients with head and neck cancer who receive radiotherapy in the United Kingdom - a web-based survey. Oral Oncol. 2012 Apr;48(4):343-8. doi: 10.1016/j.oraloncology.2011.11.003. Epub 2011 Nov 29. PMID 22130454
- [Background] McEwen S, Rodriguez AM, Martino R, Poon I, Dunphy C, Rios JN, Ringash J. "I didn't actually know there was such a thing as rehab": survivor, family, and clinician perceptions of rehabilitation following treatment for head and neck cancer. Support Care Cancer. 2016 Apr;24(4):1449-53. doi: 10.1007/s00520-015-3021-1. Epub 2015 Nov 18. PMID 26576966
- [Background] Martino R, Beaton D, Diamant NE. Using different perspectives to generate items for a new scale measuring medical outcomes of dysphagia (MOD). J Clin Epidemiol. 2009 May;62(5):518-26. doi: 10.1016/j.jclinepi.2008.05.007. Epub 2008 Aug 22. PMID 18722085
- [Background] Nund RL, Ward EC, Scarinci NA, Cartmill B, Kuipers P, Porceddu SV. Carers' experiences of dysphagia in people treated for head and neck cancer: a qualitative study. Dysphagia. 2014 Aug;29(4):450-8. doi: 10.1007/s00455-014-9527-8. Epub 2014 May 21. PMID 24844768
- [Background] List MA, Mumby P, Haraf D, Siston A, Mick R, MacCracken E, Vokes E. Performance and quality of life outcome in patients completing concomitant chemoradiotherapy protocols for head and neck cancer. Qual Life Res. 1997 Apr;6(3):274-84. doi: 10.1023/a:1026419023481. PMID 9226985
- [Background] Chen AY, Frankowski R, Bishop-Leone J, Hebert T, Leyk S, Lewin J, Goepfert H. The development and validation of a dysphagia-specific quality-of-life questionnaire for patients with head and neck cancer: the M. D. Anderson dysphagia inventory. Arch Otolaryngol Head Neck Surg. 2001 Jul;127(7):870-6. PMID 11448365
- [Background] Rosenthal DI, Mendoza TR, Chambers MS, Asper JA, Gning I, Kies MS, Weber RS, Lewin JS, Garden AS, Ang KK, S Wang X, Cleeland CS. Measuring head and neck cancer symptom burden: the development and validation of the M. D. Anderson symptom inventory, head and neck module. Head Neck. 2007 Oct;29(10):923-31. doi: 10.1002/hed.20602. PMID 17358040
- [Background] Cleeland CS, Mendoza TR, Wang XS, Chou C, Harle MT, Morrissey M, Engstrom MC. Assessing symptom distress in cancer patients: the M.D. Anderson Symptom Inventory. Cancer. 2000 Oct 1;89(7):1634-46. doi: 10.1002/1097-0142(20001001)89:73.0.co;2-v. PMID 11013380
- [Background] Martino R, Ringash J, Durkin L, Greco E, Huang SH, Xu W, Longo CJ. Feasibility of assessing patient health benefits and incurred costs resulting from early dysphagia intervention during and immediately after chemoradiotherapy for head-and-neck cancer. Curr Oncol. 2017 Dec;24(6):e466-e476. doi: 10.3747/co.24.3543. Epub 2017 Dec 20. PMID 29270055
- [Background] Greco E, Simic T, Ringash J, Tomlinson G, Inamoto Y, Martino R. Dysphagia Treatment for Patients With Head and Neck Cancer Undergoing Radiation Therapy: A Meta-analysis Review. Int J Radiat Oncol Biol Phys. 2018 Jun 1;101(2):421-444. doi: 10.1016/j.ijrobp.2018.01.097. Epub 2018 Feb 6. PMID 29726363
- [Derived] Martino R, Fitch MI, Fuller CD, Hope A, Krisciunas G, Langmore SE, Lazarus C, Macdonald CL, McCulloch T, Mills G, Palma DA, Pytynia K, Ringash J, Sultanem K, Theurer J, Thorpe KE, Hutcheson K. The PRO-ACTIVE trial protocol: a randomized study comparing the effectiveness of PROphylACTic swallow InterVEntion for patients receiving radiotherapy for head and neck cancer. BMC Cancer. 2021 Oct 13;21(1):1100. doi: 10.1186/s12885-021-08826-0. PMID 34645411